CLINICAL TRIAL: NCT05376215
Title: A Comparison of Hearing Aid Fitting Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SRF-1236
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: This study is a prospective, repeated measures, within-subject, cross over design. Subjects will be assigned in random order to the two fitting methods. Subjects will be blinded as to which fitting method they are using during the home trials.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be fit with two sets of identical devices. One set will be programmed to fitting method A and one set will be programmed to fitting method B. Subjects will be blinded as to which set they are sent on a home trial with. Outcomes will be assessed at return visits by a second sub-investigator who does not know which devices the subject is wearing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fitting method A first, then fitting method B (Active Comparator): Participants will be fit with a set of hearing devices that are programmed to fitting method A first. This fitting method will use specific programming parameters and software to determine the most appropriate fitting algorithm.
  Following a home trial with fitting method A, participants will then be fit with a set of hearing devices that are programmed to fitting method B. This fitting method will use a different set of programming parameters and software to determine the most appropriate algorithm.
  Interventions: Device: Experimental hearing aid
- Fitting method B first, then fitting method A (Experimental): Participants will be fit with a set of hearing aids that are programmed using fitting method B. This fitting method will use a different set of programming parameters and software to determine the most appropriate algorithm.
  Following a home trial with fitting method B, participants will then be fit with a set of hearing devices that are programmed to fitting method A. This fitting method will use specific programming parameters and software to determine the most appropriate fitting algorithm.
  Interventions: Device: Experimental hearing aid

INTERVENTIONS:
Device: Experimental hearing aid — This hearing aid is a receiver-in-canal style hearing aid which can be programmed and adjusted by proprietary software and by use with a mobile application.

SUMMARY:
This investigation will compare hearing aid fitting methods between self-fitting and clinician fitting approaches by using a standardized questionnaire to evaluate subjective hearing aid benefit.

DETAILED DESCRIPTION:
Participants will be fit with hearing aids using two different fitting methods (fitting A and fitting B). The order of the fitting will be randomized such that half of the participants will start out with fitting A and half of the participants will start out with fitting B. All participants will undergo baseline speech testing and answer a questionnaire about their experiences in daily life without hearing aids. All participants will use devices for a period of 1-2 weeks in their daily lives. After this first home trial, participants will return to the clinic where they will answer questionnaires regarding their experience with the devices. They will also perform aided speech testing. They will then be given devices with the second fitting method and will wear devices for a period of 1-2 weeks in their daily lives. Following the second home trial, all participants will return to the clinic to answer the same questionnaire that was given after home trial #1, and complete aided speech testing. The results for each of the two fitting methods will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate bilateral hearing loss
* First time (new) hearing aid users or experienced hearing aid users
* Ability to use a smartphone
* Fluent in English; ability to read and write in English
* Willing and able to provide informed consent

Exclusion Criteria:

* Self reported ear-related pathology including otorrhea within 90 days, dizziness, sudden onset or worsening of hearing loss within 90 days, visible deformity of the ear, otalgia
* Unilateral hearing loss
* Chronic, severe tinnitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the initial appointment in which participants were fit with both fitting methods, there was a wash out period of 1-5 days. After the wash-out period, participants returned to the site at which time they were assigned/randomized into an arm of the study. This wash-out period provided time to reduce the possibility that participants would remember how each fitting method sounded to them, and therefore reduce the chance for bias.
Groups:
- Fitting Method A First, Then Fitting Method B: Participants will be fit with a set of hearing devices that are programmed to fitting method A first. This fitting method will use specific programming parameters and software to determine the most appropriate fitting algorithm.
  Following a home trial with fitting method A, participants will then be fit with a set of hearing devices that are programmed to fitting method B. This fitting method will use a different set of programming parameters and software to determine the most appropriate algorithm.
  Experimental hearing aid: This hearing aid is a receiver-in-canal style hearing aid which can be programmed and adjusted by proprietary software and by use with a mobile application.
- Fitting Method B First, Then Fitting Method A: Participants will be fit with a set of hearing aids that are programmed using fitting method B. This fitting method will use a different set of programming parameters and software to determine the most appropriate algorithm.
  Following a home trial with fitting method B, participants will then be fit with a set of hearing devices that are programmed to fitting method A. This fitting method will use specific programming parameters and software to determine the most appropriate fitting algorithm.
  Experimental hearing aid: This hearing aid is a receiver-in-canal style hearing aid which can be programmed and adjusted by proprietary software and by use with a mobile application.
Period: Overall Study
Arm/Group | Fitting Method A First, Then Fitting Method B | Fitting Method B First, Then Fitting Method A
Started | 23 | 21
Completed First Assigned Fitting Method | 22 | 20
Completed Second Fitting Method | 21 | 19
Completed | 21 | 19
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fitting Method A First, Then Fitting Method B | Fitting Method B First, Then Fitting Method A | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11.68) | 68 (7.94) | 68 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 14 | 11 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: A validated questionnaire that assesses the subjective benefit of hearing aids in daily life. Participants rate their difficulty hearing in different situations, going from Always (99%), Almost Always (87%), Generally (75%), Half the time (50%), Occasionally (25%), Seldom (12%) or Never (1%). For example, the participant may choose "Always" to the statement "When I am having a quiet conversation with a friend, I have difficulty understanding". The questions are categorized into 4 different sub-scales: Ease of Communication (EC), Background Noise (BN), Reverberation (RV), and Aversiveness. The global score is calculated by taking the average of three of the subscales: EC, BN, and RV. The scores can range from 1% to 99%. Global Benefit is calculated by subtracting the aided global score from the unaided global score. The mean global benefit is calculated for each fitting method, and a higher benefit score is better. Result reported is the global benefit score for each fitting method.
Time Frame: Day 1 (unaided testing), Day 14(aided testing for first fitting method) and Day 28 (aided testing for second fitting method) of study
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Fitting Method A: All participants who completed a home trial with devices using fitting method A.
- Fitting Method B: All participants who completed a home trial with devices using fitting method B.
Arm/Group | Fitting Method A | Fitting Method B
Number analyzed (Participants) | 41 | 41
score on a scale | 0.099 (0.1695) | 0.106 (0.1309)
Statistical Analysis 1: Comparison: Fitting Method A vs Fitting Method B; Test type: Non-Inferiority — The non-inferiority margin of -12.5 was used per the findings from Chisolm, et al (2005), see attached article. In that study, the smallest critical difference for the short term retest difference was 12.5 for the APHAB global score at the 90th percentile. For this study, non-inferiority is confirmed if Fitting Method B is no more than 12.5 percentage points below the mean global benefit score of Fitting Method A; p = 0.806, Mixed Models Analysis

2. Secondary Outcome: Speech Perception in Noise, Expressed in Decibel (dB) Signal to Noise Ratio (SNR) Loss
Description: Objective speech in noise testing calculates the level in which speech stimuli needs to be louder than background noise for the participant to correctly repeat back 50% of key words. A lower score/dB level is better. For example, a score of 2 dB means that the speech needs to be louder than the background noise by 2 dB in order for the individual to correctly repeat 50% of the words. However, a score of 10 dB means that the speech needs to be 10 dB louder than the background noise for the individual to correctly repeat 50% of the words. This test is done in the unaided condition, as well as with both aided conditions (fitting method A and fitting method B) and the benefit score for each fitting method is determined by subtracting the aided dB SNR score from the unaided dB SNR score. A higher benefit score is better.
Time Frame: Day 1 (unaided/baseline testing) of study, day 14 (aided testing with first fitting method) and day 28 (aided testing with second fitting method) of study
Population: All participants who completed unaided/baseline speech in noise testing and aided speech in noise testing with both fitting methods so that the aided benefit score could be calculated.
Measure: Mean (Standard Deviation); unit: decibels (dB)
Arm/Group | Fitting Method A | Fitting Method B
Number analyzed (Participants) | 40 | 40
decibels (dB) | -0.131 (1.81) | -0.069 (1.54)
Statistical Analysis 1: Comparison: Fitting Method A vs Fitting Method B; Test type: Non-Inferiority — The non-inferiority margin is -1.8 dB. This is based off of work by Killion (2004) in which the critical difference for 4 lists is 1.9 dB at the 95% confidence interval. Killion also found that if all 12 lists are presented, the mean SNR scores will differ by 1.8 dB 5% of the time; p = 0.889, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Four weeks
Groups:
- Fitting Method A: All enrolled participants who completed a two week home trial with Fitting Method A.
  Experimental hearing aid: This hearing aid is a receiver-in-canal style hearing aid which can be programmed and adjusted by proprietary software and by use with a mobile application.
- Fitting Method B: All enrolled participants who completed a two week home trial with Fitting Method B.
  Experimental hearing aid: This hearing aid is a receiver-in-canal style hearing aid which can be programmed and adjusted by proprietary software and by use with a mobile application.
Arm/Group | Fitting Method A | Fitting Method B
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 1/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fitting Method A (N=41) | Fitting Method B (N=41)
ear canal occlusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Plugged and occluded sensation in ear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to any publication or presentation, Sonova reserves the right to review, oppose, or restrict the publication or presentation of protected intellectual property and/or confidential information. If an objection is raised by Sonova, discussion shall be held without delay to determine acceptable modifications to resolve the issue and allow dissemination within sixty days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT05376215/Prot_SAP_000.pdf